CLINICAL TRIAL: NCT06189781
Title: Peri-operative Use of a Pain Injection Versus Epidural in Pediatric Patients With Cerebral Palsy
Brief Title: Pain Injection Versus Epidural Anesthesia for Hip Surgery in Pediatric Patients With Cerebral Palsy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Rachel Thompson, MD, Director, Center for Cerebral Palsy, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#23-000902
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy; Hip Dysplasia; Pain, Postoperative
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation; Pain, Postoperative | interventions — Ropivacaine; Bupivacaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to either treatment/intervention group (injection only) or control (epidural only). All other aspects of care will be identical between the two groups.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Injection (Experimental): The local anesthetic group will be injected with a combination of ropivacaine, epinephrine, and ketorolac.
  Interventions: Drug: Ropivacaine injection
- Epidural (Active Comparator): The control group will receive epidural anesthesia. Lumbar epidural anesthesia will be started intra-operatively.
  Interventions: Drug: Bupivacaine, lidocaine, ropivacaine

INTERVENTIONS:
Drug: Ropivacaine injection — The local anesthetic group will be injected with ropivacaine 2mg/mL (3mg/kg), epinephrine 1mg/mL (0.5mg), and ketorolac 30mg/mL (0.5mg/kg). The maximum dose of ropivacaine regardless of patient weight will be 200mg. This is based on recommended maximum dose protocols from our anesthesia colleagues. If bilateral hips are involved, the total amount will be split evenly between the two sides.
  Arms: Pain Injection
Drug: Bupivacaine, lidocaine, ropivacaine — The lumbar epidural group will receive a combination of either/or bupivacaine, lidocaine, and ropivacaine, which will be monitored by the anesthesia team.
  Arms: Epidural

SUMMARY:
Pain management in pediatric patients presents a difficult challenge. Unlike adults, pediatric patients often cannot communicate their pain management needs clearly. This is especially true in patients with cerebral palsy (CP), who often have concomitant developmental delay, intellectual disability and verbal limitations. Current literature indicates pain as a common experience for children with CP but has been understudied in this population. Moreover, inadequate post-operative pain control can result in negative physiologic and psychological complications and lead to poor surgical outcomes. Currently, perioperative pain management following orthopaedic procedures in pediatric patients follows traditional protocols that rely on the administration of opioid medications despite their known adverse side effects including nausea, vomiting, itching, constipation, urinary retention, confusion, and respiratory depression.

Epidural anesthesia is a key modality in traditional pain management for pediatric patients with CP given its proven efficacy in decreasing pain and managing spasticity. Yet, administering epidural anesthesia in this patient population poses several risks including damage to preexisting intrathecal baclofen pumps, iatrogenic infection, and technically demanding insertion given high rates of concomitant neuromuscular scoliosis. Alternatively, multimodal analgesic injections theoretically offer an efficacious adjunct to traditional pain management protocols with a lower risk profile. Preliminary data from our study group's pilot randomized control trial comparing the safety and efficacy of a multimodal surgical site injection to placebo showed decreased pain scores and narcotic consumption postoperatively in this patient population. Based on these promising results, the objective of this randomized control trial is to evaluate the efficacy of a multimodal surgical site injection compared to epidural anesthesia for postoperative pain control following operative management of hip dysplasia in pediatric patients with CP.

DETAILED DESCRIPTION:
Over the past decade, there has been an ongoing shift away from the use of opioids in the postoperative setting due to both their negative side effects and their high potential for dependence and abuse. Various new techniques for multimodal pain management are increasingly being utilized in adult orthopaedics, including injection of local anesthetics and analgesic agents. These techniques aim to block pain directly at the site of injection in order to reduce postoperative pain while minimizing systemic effects and preserving motor function, allowing for early mobilization. Numerous randomized controlled trials in both the arthroplasty and adult trauma populations have demonstrated reduced pain and narcotic consumption with local analgesia injection, but there is scant evidence on the efficacy of similar injections in pediatric surgical patients. While robust evidence demonstrating both safety and efficacy of these injections has led to routine use in the adult orthopaedic population, use in pediatric patients still remains limited, likely due to a lack of level I therapeutic evidence.

Local anesthetic injections offer several theoretical advantages over current pain management modalities. When compared with other methods of anesthesia, including epidural anesthesia or some peripheral nerve blocks, local anesthetic injections preserve motor function, allowing for early mobilization and rehabilitation. Additionally, they do not require specialized equipment or anesthesia personnel and can be administered in the operating room without significantly affecting the duration of the procedure. While a mainstay in traditional pain management protocols, epidural anesthesia in the pediatric CP population poses specific risks including damage to preexisting intrathecal baclofen pumps and iatrogenic infection. Moreover, epidural insertion can be a technically demanding procedure in these patients given high rates of concomitant neuromuscular scoliosis. Prior retrospective studies comparing peripheral nerve and lumbar plexus blocks compared to epidural anesthesia have shown mixed results in decreasing pain scores and opioid use in this patient population. As described in Preliminary Data section below, the investigators' pilot randomized control trial demonstrated significantly decreased pain scores and narcotic use postoperatively in pediatric patients with CP who received multimodal analgesia injection compared to placebo while undergoing hip surgery. The present study aims to substantively contribute to current literature by providing level I evidence comparing the safety and efficacy of surgical site injections with epidural anesthesia in a patient population for whom pain management remains challenging.

ELIGIBILITY:
Inclusion Criteria:

* under 18 years old
* diagnosis of cerebral palsy or similar neuromuscular disease
* undergoing uni- or bilateral proximal femoral osteotomy

Exclusion Criteria:

* ongoing preoperative opioid use
* history of allergic reaction to any component of the pain injection
* history of adverse reaction to epidural anesthesia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Average postoperative narcotic consumption measured in morphine equivalents per kilograms of patient body weight | First 48 hours after surgery
  This describes one outcome measure where the amount of opiates consumed will be expressed in morphine equivalents divided by the body weight of patients measured in kilograms.

SECONDARY OUTCOMES:
Postoperative pain scores measured by Visual Analogue Scale/Faces Pain Scale/Face, Legs, Activity, Cry, Consolability Scale | 2-4 days
  Pain score assessments will be completed in the post-anesthesia care unit, and every 4 hours following the surgical procedure. Scores will be collected by nursing staff on the inpatient ward and recorded in the electronic medical record. The type of pain score collection will vary based on patient age and level of intellectual disability. In verbal children, either the Visual Analogue Scale or Faces Pain Scale will be employed. In non-verbal children, the Face, Legs, Activity, Cry, Consolability Scale will be employed. A higher score indicates greater pain intensity. Both scales are from 0 (minimum) -10 (maximum), where 0 indicates no pain and 10 indicate maximal pain.
Hospital length of stay measured in days | 2-4 days
  Postoperative hospital length of stay
Parent satisfaction measured on a scale of 1-5 | 2-3 weeks postoperatively
  Parent satisfaction will be based on a standardized, validated questionnaire taken by parents in person at the first post-operative clinic visit aimed to assess their satisfaction with their child's pain management peri-operatively. Each question is answered with a score of either 1-5, with 1 being the best outcome and 5 being the worst outcome. The score for each question will be summed together to come up with a total score. A higher total score indicates a worse level of satisfaction with perioperative pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Thompson, MD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - Orthopaedic Institute for Children, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson KB, Emery ES 3rd. Birth asphyxia and the neonatal brain: what do we know and when do we know it? Clin Perinatol. 1993 Jun;20(2):327-44. PMID 8358954
- [Background] Nolan J, Chalkiadis GA, Low J, Olesch CA, Brown TC. Anaesthesia and pain management in cerebral palsy. Anaesthesia. 2000 Jan;55(1):32-41. doi: 10.1046/j.1365-2044.2000.01065.x. PMID 10594431
- [Background] Tabaie S, Shah A, Tarawneh O, Blaylock G, Sheppard E, Cho K. Use of Epidural Analgesia in Children With Neuromuscular Conditions Following Hip Reconstruction. Cureus. 2022 Oct 20;14(10):e30522. doi: 10.7759/cureus.30522. eCollection 2022 Oct. PMID 36285108
- [Background] Hauer J, Houtrow AJ; SECTION ON HOSPICE AND PALLIATIVE MEDICINE, COUNCIL ON CHILDREN WITH DISABILITIES. Pain Assessment and Treatment in Children With Significant Impairment of the Central Nervous System. Pediatrics. 2017 Jun;139(6):e20171002. doi: 10.1542/peds.2017-1002. PMID 28562301
- [Background] McKearnan KA, Kieckhefer GM, Engel JM, Jensen MP, Labyak S. Pain in children with cerebral palsy: a review. J Neurosci Nurs. 2004 Oct;36(5):252-9. doi: 10.1097/01376517-200410000-00004. PMID 15524243
- [Background] Ciccozzi A, Pizzi B, Vittori A, Piroli A, Marrocco G, Della Vecchia F, Cascella M, Petrucci E, Marinangeli F. The Perioperative Anesthetic Management of the Pediatric Patient with Special Needs: An Overview of Literature. Children (Basel). 2022 Sep 21;9(10):1438. doi: 10.3390/children9101438. PMID 36291372
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Piper NA, Flack SH, Loeser JD, Lynn AM. Epidural analgesia in a patient with an intrathecal catheter and subcutaneous pump to deliver baclofen. Paediatr Anaesth. 2006 Sep;16(9):989-92. doi: 10.1111/j.1460-9592.2006.01908.x. PMID 16918665
- [Background] Fiore JF Jr, Olleik G, El-Kefraoui C, Verdolin B, Kouyoumdjian A, Alldrit A, Figueiredo AG, Valanci S, Marquez-GdeV JA, Schulz M, Moldoveanu D, Nguyen-Powanda P, Best G, Banks A, Landry T, Pecorelli N, Baldini G, Feldman LS. Preventing opioid prescription after major surgery: a scoping review of opioid-free analgesia. Br J Anaesth. 2019 Nov;123(5):627-636. doi: 10.1016/j.bja.2019.08.014. Epub 2019 Sep 25. PMID 31563269
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Background] Peters CL, Shirley B, Erickson J. The effect of a new multimodal perioperative anesthetic regimen on postoperative pain, side effects, rehabilitation, and length of hospital stay after total joint arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):132-8. doi: 10.1016/j.arth.2006.04.017. PMID 16950075
- [Background] Andersen KV, Pfeiffer-Jensen M, Haraldsted V, Soballe K. Reduced hospital stay and narcotic consumption, and improved mobilization with local and intraarticular infiltration after hip arthroplasty: a randomized clinical trial of an intraarticular technique versus epidural infusion in 80 patients. Acta Orthop. 2007 Apr;78(2):180-6. doi: 10.1080/17453670710013654. PMID 17464604
- [Background] Koehler D, Marsh JL, Karam M, Fruehling C, Willey M. Efficacy of Surgical-Site, Multimodal Drug Injection Following Operative Management of Femoral Fractures: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Mar 15;99(6):512-519. doi: 10.2106/JBJS.16.00733. PMID 28291185
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Uesugi K, Kitano N, Kikuchi T, Sekiguchi M, Konno S. Comparison of peripheral nerve block with periarticular injection analgesia after total knee arthroplasty: a randomized, controlled study. Knee. 2014 Aug;21(4):848-52. doi: 10.1016/j.knee.2014.04.008. Epub 2014 Apr 18. PMID 24827696
- [Background] Laron D, Kelley J, Chidambaran V, McCarthy J. Fascia Iliaca Pain Block Results in Lower Overall Opioid Usage and Shorter Hospital Stays than Epidural Anesthesia After Hip Reconstruction in Children With Cerebral Palsy. J Pediatr Orthop. 2022 Feb 1;42(2):96-99. doi: 10.1097/BPO.0000000000002028. PMID 34882587